CLINICAL TRIAL: NCT03403426
Title: A Non-Randomized Study Evaluating the Use of the ReFlow Medical Wingman Catheter to Cross Chronic Total Occlusions in Infrainguinal Peripheral ArTeries
Brief Title: ReFlow Medical Wingman Catheter Wing-IT Clinical Trial
Acronym: Wing-It
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ReFlow Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RFM-CTO-13001
Record Dates: First submitted 2017-11-29; First posted 2018-01-18 (Actual); Results first posted 2021-01-07 (Actual); Last update posted 2021-01-07 (Actual); Status verified 2021-01

CONDITIONS: Chronic Total Occlusion of Artery of the Extremities

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Wingman Crossing Catheter (Experimental): Use of the device to support CTO crossing
  Interventions: Device: Wingman Crossing Catheter

INTERVENTIONS:
Device: Wingman Crossing Catheter — Endovascular CTO crossing

SUMMARY:
To evaluate the safety and effectiveness of the ReFlow Medical Wingman Catheter used to cross de novo or restenotic infrainguinal CTOs that cannot be crossed with a standard guidewire.

DETAILED DESCRIPTION:
Prospective, multi-center, non-randomized single-arm study of the Wingman Catheter to cross a single infrainguinal peripheral chronic total occlusion (CTO). Safety and effectiveness will be evaluated during the index procedure through 30-day follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patient is willing and able to provide informed consent.
* Patient is willing and able to comply with the study protocol.
* Patient is > 18 years old.
* Patient has peripheral arterial disease requiring revascularization as evidenced by contrast, CT or MR angiography.
* Patient has at least one but not more than two occluded infrainguinal arteries that are 99-100% stenosed and no flow is observed in the distal lesion except the flow from collateral circulation.
* Target lesion(s) is ≥ 1 cm and < 30 cm in length by visual estimate.
* Target vessel is ≥ 2.0 mm in diameter.
* Patient has Rutherford Classification of 2-5.
* Lesion cannot be crossed by concurrent conventional guidewire.
* Reconstitution of vessel at least 2cm above bifurcation/trifurcation.
* Occlusion can be within previously implanted stent.

Exclusion Criteria:

* Patient has a known sensitivity or allergy to contrast materials that cannot be adequately pre-treated.
* Patient has a known sensitivity or allergy to all anti-platelet medications.
* Patient is pregnant or lactating.
* Patient has a co-existing disease or medical condition contraindicating percutaneous intervention.
* Target lesion is in a bypass graft.
* Patient has had a failed crossing attempt without an intervening intervention on the target limb within the past 14 days.
* Patient has a planned surgical or interventional procedure within 30 days after the study procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2018-02-13 (Actual); Primary Completion 2019-08-08 (Actual); Study Completion 2019-08-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Laird, MD, Principal Investigator — Adventist St. Helena Hospital
Locations (1):
- Adventist St. Helena Hospital, St. Helena, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Wingman Crossing Catheter
Started | 85
Completed | 82
Not Completed | 3
Not completed — Death | 1
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Units Other Than Participants: lesions
Arm/Group | Wingman Crossing Catheter
Number analyzed (Participants) | 85
Number analyzed (lesions) | 86
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.4 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 56
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 84
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 78
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 59
  Austria | 15
  Germany | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Lesions With Successful CTO Crossing Assessed by Angiography
Description: While using the Wingman device, successful CTO crossing is identified by successful guidewire placement in the distal true lumen confirmed by angiography with no clinically significant perforations. Assessment by angiography with results reviewed by an independent core lab.
Time Frame: Intraprocedural
Measure: Count of Units; unit: lesions
Units Other Than Participants: lesions
Arm/Group | Wingman Crossing Catheter
Number analyzed (Participants) | 85
Number analyzed (lesions) | 86
lesions | 77

2. Primary Outcome: Major Adverse Event (MAE) Rate
Description: Occurrence of significant in-hospital or 30-day MAEs.
Time Frame: Assessed from the time of the procedure through 30 days
Population: Denominator is not to equal to 85 due to incomplete 30-day follow-up data. 1 subject was lost to follow-up and 1 subject withdrew after 30 days but did not have a 30 day visit.
  All 85 patients were monitored for AEs in-hospital, but as the primary endpoint is through 30 days 2 of the patients were not included in the analysis after they withdrew or were lost to follow-up. Any adverse events were captured and reported in the adverse event module for all 85 patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Wingman Crossing Catheter
Number analyzed (Participants) | 83
Participants | 4

3. Primary Outcome: Rate of Clinically Significant Perforations
Description: Occurrence of clinically significant perforation, after Wingman CTO crossing and PTA of lesion, confirmed by angiography, evaluated by angiographic core lab
Time Frame: Will be assessed from the time of the procedure through 30 days
Population: Denominator is not to equal to 85 due to incomplete 30-day follow-up data. 1 subject was lost to follow-up and 1 subject withdrew after 30 days but did not have a 30 day visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Wingman Crossing Catheter
Number analyzed (Participants) | 83
Participants | 1

4. Secondary Outcome: Lesion Success
Description: Lesion success, defined as attainment of <50% final residual stenosis of the target lesion using any percutaneous method
Time Frame: Intraprocedural
Population: Denominator is not equal to 86 lesion due to missing data points in 3 patients.
Measure: Count of Units; unit: Lesions
Units Other Than Participants: Lesions
Arm/Group | Wingman Crossing Catheter
Number analyzed (Participants) | 85
Number analyzed (Lesions) | 83
Lesions | 77

5. Secondary Outcome: Procedure Success Rate
Description: Procedure success, defined as device success and the absence of in-hospital MAEs, clinically significant perforation, clinically significant embolization or Grade C or greater dissection not resolved by visual estimate
Time Frame: Approximately 24 hours post procedure
Population: Denominator is not to equal to 85 due to missing data points on 3 subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Wingman Crossing Catheter
Number analyzed (Participants) | 82
Participants | 75

6. Secondary Outcome: Incidence of In-hospital AE or MAE
Description: Procedure safety defined as any in-hospital AE or MAE following use of a therapeutic interventional device
Time Frame: Intraprocedural
Measure: Count of Participants; unit: Participants
Arm/Group | Wingman Crossing Catheter
Number analyzed (Participants) | 85
Participants | 16

7. Secondary Outcome: Total Procedural Time
Description: Evaluation of total procedural time
Time Frame: Approximately 24 hours post procedure
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Wingman Crossing Catheter
Number analyzed (Participants) | 85
minutes | 102 (48)

8. Secondary Outcome: Device Procedural Time
Description: Evaluation of procedure time associated with use of the investigational device.
Time Frame: Approximately 24 hours post procedure
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Wingman Crossing Catheter
Number analyzed (Participants) | 85
minutes | 12 (12)

9. Secondary Outcome: Contrast Use
Description: Evaluation of total procedural contrast volume use
Time Frame: Approximately 24 hours post procedure
Population: Denominator is not to equal to 85 due to missing data on 4 patients.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Wingman Crossing Catheter
Number analyzed (Participants) | 81
mL | 148 (79)

10. Secondary Outcome: Fluoroscopic Time
Description: Evaluation of total procedural fluoroscopic time
Time Frame: Approximately 24 hours post procedure
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Wingman Crossing Catheter
Number analyzed (Participants) | 85
minutes | 30 (18)

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Wingman Crossing Catheter
All-Cause Mortality (participants affected / at risk) | 1/85
Serious Adverse Events (participants affected / at risk) | 22/85
Other Adverse Events (participants affected / at risk) | 21/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Wingman Crossing Catheter (N=85)
Acute left ventricular failure (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Ventricular fibrillation (Cardiac disorders) | 1
Procedural vomiting (Gastrointestinal disorders) | 1
Vascular stent occlusion (General disorders) | 1
Vascular access site pain (General disorders) | 1
Vascular access site dissection (General disorders) | 2
Arterial perforation (General disorders) | 1
Vascular access site pseudoaneurysm (General disorders) | 1
Contrast media reaction (Immune system disorders) | 1
Gangrene (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Abscess limb (Infections and infestations) | 1
Vascular access site haematoma (Injury, poisoning and procedural complications) | 1
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 3
Arterial bypass thrombosis (Injury, poisoning and procedural complications) | 1
Vessel perforation (Injury, poisoning and procedural complications) | 2
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1
Respiratory failure (Metabolism and nutrition disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Subclavian steal syndrome (Nervous system disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1
Arteriovenous fistula (Vascular disorders) | 1
Peripheral embolism (Vascular disorders) | 1
Peripheral artery thrombosis (Vascular disorders) | 1
Peripheral artery occlusion (Vascular disorders) | 4
Intermittent claudication (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Wingman Crossing Catheter (N=85)
Vascular access site dissection (General disorders) | 10
Vascular access site haematoma (General disorders) | 7
Peripheral embolism (Vascular disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-05-20): https://cdn.clinicaltrials.gov/large-docs/26/NCT03403426/SAP_000.pdf
  • Study Protocol (2018-10-03): https://cdn.clinicaltrials.gov/large-docs/26/NCT03403426/Prot_001.pdf